CLINICAL TRIAL: NCT00225563
Title: Transforming Healthcare Quality Through I.T.
Brief Title: Taconic Health Information Network and Community (THINC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 7UC1HS015316-02 (AHRQ)
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2018-06

CONDITIONS: Medication Errors
Keywords: Electronic medical records; Electronic prescribing; Quality measures
MeSH Terms: interventions — Electronic Health Records

STUDY DESIGN:
Intervention Model Description: The study model used pre-post design of 15 providers who adopted e-prescribing with concurrent controls of 15 paper-based providers from September 2005 through June 2007.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-prescribing (Active Comparator): Providers who used electronic prescriptions. electronic health records were used as opposed to paper based prescriptions
  Interventions: Device: Electronic Health Record
- Paper-based prescriptions (No Intervention): providers who used paper based prescriptions

INTERVENTIONS:
Device: Electronic Health Record — e-prescribing methods
  Arms: e-prescribing

SUMMARY:
The Taconic IPA, a 2,500 physician independent practice association (IPA) located in Fishkill, New York (NY), is involved in an information technology project to improve the quality, safety and efficiency of healthcare in the region. Over the past three years, the organization has worked with area hospitals and laboratories to create a community wide electronic data exchange. Currently, the Taconic IPA is in the midst of implementing a full electronic health record in some practices and e-prescribing in other practices. The purpose is to study the impact of an electronic health record on safety and quality measures.

DETAILED DESCRIPTION:
We propose to measure differences in patient safety and quality measures among three groups: the control group consisting of physicians with paper-based office practices, a group of physicians using the clinical messaging system and electronic prescribing, and a group of physicians using the EMR and electronic prescribing.

We plan to introduce a vendor based electronic prescribing system by July 2005. This system will be offered to all physicians using clinical messaging and will be integrated with the EMR system. The system will have clinical decision support, such as checks for drug-drug interactions.

Our evaluation will measure differences in rates of medication errors and quality measures amongst these three groups. We will use a study design of a pre-post evaluation with a comparison control group. We will detect medical errors by prescription and chart review. We will determine compliance with quality measures through a combination of electronic data and chart review.

ELIGIBILITY:
Inclusion Criteria:

* Physicians' prescriptions and medical records in office practices enrolled in the study

Exclusion Criteria:

* Other physicians not enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-07-21 (Actual); Primary Completion 2012-05-25 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Medication errors | 2007-2012
Near misses | 2007-2012
Adverse drug events | 2007-2012
Quality measures | 2007-2012

CONTACTS AND LOCATIONS:
Overall Officials: A. John Blair, MD, Principal Investigator — Taconic IPA; Rainu Kaushal, MD, Principal Investigator — Partners Health Care
Locations (1):
- Taconic IPA, Fishkill, New York, United States

IPD SHARING:
Plan to Share IPD: No
not applicable. no plan to share IPD

REFERENCES:
- [Derived] Abramson EL, Barron Y, Quaresimo J, Kaushal R. Electronic prescribing within an electronic health record reduces ambulatory prescribing errors. Jt Comm J Qual Patient Saf. 2011 Oct;37(10):470-8. doi: 10.1016/s1553-7250(11)37060-2. PMID 22013821
- [Derived] Kaushal R, Kern LM, Barron Y, Quaresimo J, Abramson EL. Electronic prescribing improves medication safety in community-based office practices. J Gen Intern Med. 2010 Jun;25(6):530-6. doi: 10.1007/s11606-009-1238-8. Epub 2010 Feb 26. PMID 20186499